CLINICAL TRIAL: NCT00348569
Title: A Prospective, Multicenter Study of GE LightSpeed Volume Computed Tomography (CT) for Evaluation of Coronary Artery Blockages in Typical or Atypical Chest Pain Patients Suspected of Coronary Artery Disease
Brief Title: A Study of Computed Tomography (CT) for Evaluation of Coronary Artery Blockages in Typical or Atypical Chest Pain
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: GE Healthcare (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: GE-189-002
Record Dates: First submitted 2006-06-30; First posted 2006-07-04 (Estimated); Last update posted 2019-04-29 (Actual); Status verified 2019-04

CONDITIONS: Coronary Artery Disease
Keywords: CT; Coronary; Cardiac; Angiography; X-ray; CAD; Chest pain
MeSH Terms: conditions — Coronary Artery Disease; Chest Pain

ARMS (1):
- 64 Channel VCT (Experimental): All subjects underwent Coronary Computed Tomographic Angiography (CCTA) after receiving an intravenous (IV) administration of Visipaque (320 mgI/mL), to be followed 2 to 21 days later by catheter coronary angiography (CATH).
  Interventions: Device: 64 Channel VCT

INTERVENTIONS:
Device: 64 Channel VCT

SUMMARY:
To compare computed tomography (CT) images (pictures) of the coronary arteries using the General Electric (GE) LightSpeed VCT scanner with x-ray coronary angiography in patients with typical or atypical chest pain suspected of coronary artery disease (CAD).

ELIGIBILITY:
Inclusion Criteria:

* The subject has typical or atypical chest pain suspected of CAD and is referred for an elective coronary angiography.
* The subject must be scheduled to undergo a CATH procedure between 48 hours and 3 weeks post CCTA procedure.
* The subject must not undergo any cardiac interventional treatment between the 2 procedures.
* The subject must have sinus rhythm with stable heart rate of ≤65 beats per minute (bpm) or if heart rate was >65 bpm, the subject must agree to the use of beta-blocker(s) prior to the CT scan procedure to achieve stable heart rate of ≤65 bpm.

Exclusion Criteria:

* The subject had an established diagnosis of CAD by a) previous CATH, b) prior myocardial infarction confirmed by ECG, or c) prior revascularization (balloon angioplasty, stent placement, or CABG).
* The subject had a known allergy to iodinated contrast agent, including but not limited to hives, anaphylactoid or cardiovascular reactions, laryngeal edema and bronchospasm.
* The subject had impaired renal function with a serum creatinine level of 1.7 mg/dL (150 μmol/L) or above.
* The subject had atrial fibrillation/flutter or any irregular heart rhythm considered by the investigator to interfere with temporal acquisition of cardiac CT images.
* The subject had a resting heart rate of >100 bpm and/or a resting systolic blood pressure of <100mm Hg.
* The subject had an artificial heart valve(s).
* The subject has had prior pacemaker or internal defibrillator lead implantation.
* The subject's resting heart rate was >65 bpm and beta-blocker therapy was contraindicated.
* The subject had a contraindication to verapamil when beta-blocker therapy could not be administered. The subject had a contraindication to nitroglycerin.
* The subject had evidence of ongoing or active clinical instability.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 245 (Actual)
Dates: Start 2006-05; Primary Completion 2007-01-31 (Actual); Study Completion 2007-01-31 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Robert Centofanti, MS, Study Director — GE Healthcare
Locations (1):
- Robert Centofanti, MS, Princeton, New Jersey, United States

REFERENCES:
- [Derived] Min JK, Edwardes M, Lin FY, Labounty T, Weinsaft JW, Choi JH, Delago A, Shaw LJ, Berman DS, Budoff MJ. Relationship of coronary artery plaque composition to coronary artery stenosis severity: results from the prospective multicenter ACCURACY trial. Atherosclerosis. 2011 Dec;219(2):573-8. doi: 10.1016/j.atherosclerosis.2011.05.032. Epub 2011 May 31. PMID 21696739
- [Derived] Budoff MJ, Dowe D, Jollis JG, Gitter M, Sutherland J, Halamert E, Scherer M, Bellinger R, Martin A, Benton R, Delago A, Min JK. Diagnostic performance of 64-multidetector row coronary computed tomographic angiography for evaluation of coronary artery stenosis in individuals without known coronary artery disease: results from the prospective multicenter ACCURACY (Assessment by Coronary Computed Tomographic Angiography of Individuals Undergoing Invasive Coronary Angiography) trial. J Am Coll Cardiol. 2008 Nov 18;52(21):1724-32. doi: 10.1016/j.jacc.2008.07.031. PMID 19007693